CLINICAL TRIAL: NCT03445832
Title: Pulmonary Function and Neuromuscular Disease
Acronym: PREMDEN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2017/346
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to describe the evolution of pulmonary function in 3 neuromuscular diseases : Duchenne muscular dystrophy, Werdnig-Hoffinann disease, congenital myopathy, monitored in Besançon university hospital.

ELIGIBILITY:
Inclusion Criteria:

* Neuromuscular disease
* Followed-up in Besançon University Hospital
* With at least 2 Pulmonary Function Tests previously performed

Exclusion Criteria:

* Mental deficiency
* Facial expressions disorders

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children suffering from neuromuscular diseases and followed-up in Besançon University Hospital between 2006/01/01 and the beginning of this study
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
FVC (Forced Vital Capacity) | Year 12
  Percentage of decrease of FVC sitting or lying down

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France